CLINICAL TRIAL: NCT07097909
Title: A Multi-agent Large Language Model Conversational AI for Tinnitus Management: The Fudan Tinnitus Doctor Randomised Controlled Trial
Brief Title: Efficacy and Safety of LLM-Based CBT for Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LLM-TCBT
Record Dates: First submitted 2025-07-30; First posted 2025-08-01 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLM-based Conversational CBT (FTD) (Experimental): Participants in this group will receive a 30-day self-directed intervention delivered through the Fudan Tinnitus Doctor (FTD) system, a multi-agent large language model-based conversational AI platform designed to provide tinnitus-focused cognitive behavioural therapy.
  Interventions: Other: Fudan Tinnitus Doctor (FTD) Conversational AI System
- Digital Education Control Group (Active Comparator): Participants in this group will receive static, evidence-based tinnitus education materials presented through the same digital platform, matched in format and duration to the intervention group but without interactive AI components.
  Interventions: Other: Digital Education Materials

INTERVENTIONS:
Other: Fudan Tinnitus Doctor (FTD) Conversational AI System — The FTD system will deliver personalized CBT-style dialogues including tinnitus psychoeducation, cognitive restructuring, relaxation training, sleep hygiene, and mindfulness guidance. The system will operate through a secure hospital web platform, accessible via personal devices, and will incorporate retrieval-augmented generation and safety moderation to ensure evidence-based and safe interaction.
  Arms: LLM-based Conversational CBT (FTD)
Other: Digital Education Materials — Educational modules will include information on tinnitus mechanisms, common coping strategies, and general lifestyle recommendations. The materials will be accessed via the same secure platform as the intervention group to control for exposure time and digital interface effects.
  Arms: Digital Education Control Group

SUMMARY:
Given the limited evidence on digital cognitive behavioral therapy (CBT) for chronic subjective tinnitus, particularly interventions supported by large language models (LLMs), this two-arm, 30-day randomized controlled trial will aim to evaluate the efficacy, safety, and usability of an LLM-based conversational CBT intervention compared with a digital education control. Participants with chronic subjective tinnitus will be randomly assigned to either the intervention group, which will receive daily AI-supported CBT sessions through the Fudan Tinnitus Doctor (FTD) system, or the control group, which will receive static tinnitus education materials matched for duration and platform interface. The FTD system will be powered by a multi-agent large language model and will deliver personalized CBT-style dialogues, including psychoeducation, cognitive restructuring, relaxation, and mindfulness guidance. Outcomes will include tinnitus severity, sleep quality, mood symptoms, global improvement, and user adherence and experience.

DETAILED DESCRIPTION:
Chronic subjective tinnitus is a common and often distressing auditory condition that frequently co-occurs with insomnia, anxiety, and depression. Cognitive behavioral therapy (CBT) remains the most evidence-based treatment to reduce tinnitus-related distress, but traditional face-to-face CBT is limited by accessibility, cost, and availability of trained professionals. Digital CBT interventions have demonstrated potential benefits, yet their efficacy varies, and engagement and personalization remain major challenges.

Recent advances in large language models (LLMs) have enabled the development of interactive conversational systems capable of delivering psychologically informed support. The Fudan Tinnitus Doctor (FTD) is a multi-agent conversational AI platform specifically designed to provide CBT-based tinnitus management. It integrates psychoeducation, cognitive restructuring, relaxation, and mindfulness guidance within natural language conversations. The system will be powered by a multi-agent large language model with retrieval-augmented generation (RAG) and safety moderation to ensure content validity, consistency, and user safety.

This single-centre, parallel-group, open-label randomized controlled trial will evaluate the efficacy, safety, and usability of the FTD system compared with a digital education control. Participants with chronic subjective tinnitus meeting the inclusion criteria will be randomly assigned (1:1) to either the FTD intervention group or the control group. The intervention group will receive 30 days of AI-supported CBT sessions through the secure hospital web platform, while the control group will receive static tinnitus education materials matched for platform and duration but without interactive AI components.

The primary outcome will be the change in tinnitus severity measured by the Tinnitus Handicap Inventory (THI) from baseline to Day 30. Secondary outcomes will include sleep quality (Pittsburgh Sleep Quality Index, PSQI), anxiety (GAD-2), depression (PHQ-2), and overall perceived improvement (Patient Global Impression of Change, PGIC). Exploratory outcomes will assess usability (System Usability Scale, SUS), satisfaction (Net Promoter Score, NPS), and engagement metrics.

All assessments will use validated Chinese versions of the respective questionnaires. Safety monitoring will be conducted throughout the study period. Adverse events and any AI-related performance errors will be automatically logged and reviewed by the research team.

This study will provide preliminary evidence on the efficacy and safety of an LLM-based conversational CBT system for tinnitus management, offering a scalable and patient-centered approach that could enhance accessibility and adherence in digital mental health care.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of subjective tinnitus confirmed by a qualified investigator.
2. Tinnitus duration ≥ 3 month prior to screening.
3. THI score of ≥ 18
4. Aged between 18 and 70 years
5. The ability to use a smartphone: Both groups will receive therapeutic support and disease management primarily through a mobile application or web-based platform. This requires functional ability to operate the provided software and willingness to engage with the digital intervention protocol.
6. Perceptibility: Tinnitus is present and recognizable by the participant under ordinary daily conditions (not only in quiet environments).
7. Compliance and consent: Participant is assessed by the Investigator as able to understand study procedures, voluntarily agrees to participate, is willing to comply with all trial-related requirements, and provides signed informed consent prior to performance of any protocol-specified procedure.

Exclusion Criteria:

1. Acute-phase tinnitus (duration < 3 month or tinnitus secondary to acute otologic events).
2. Pulsatile or objective tinnitus.
3. Unstable symptoms: Fluctuating tinnitus loudness at screening or baseline.
4. Psychiatric contraindication: History or current presence of severe psychiatric disorders (e.g., major depressive disorder with recent suicidality, schizophrenia) that, in the opinion of the Investigator, may interfere with study participation or data validity.
5. Testing limitations: Inability to adequately complete tinnitus testing procedures or comply with study assessments.
6. Prior therapy exposure: Previous history of sound therapy specifically for tinnitus management.
7. Concurrent treatments: Ongoing psychotherapy for conditions such as anxiety or depression, or any other psychological treatment that may interfere with the study endpoints.
8. Concurrent trial participation: Active participation in another interventional research study that, in the opinion of the Investigator, could affect tinnitus symptoms or interact with study procedures.
9. Investigator judgment: Any condition (medical, surgical, psychiatric, or social) or factor which, in the Investigator's judgment, renders the subject unsuitable for participation, places the patient at higher risk, or may interfere with compliance or scientific validity of the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2025-08-02 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | Baseline, Day 14, and Day 30
  The THI questionnaire, widely used in research, including functional, emotional, and catastrophic subscales. It consists of 25 questions, and answers are rated on a "yes" (4 points), "sometimes" (2 points), and "no" (0 points) scale. The total score is calculated by adding up the scores for all questions and classifying the severity of tinnitus as no handicap (0-16), mild handicap (18-36), moderate handicap (38-56), and severe handicap (58-100).

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Baseline, Day 14, and Day 30
  The PSQI will be used to evaluate subjective sleep quality over the past month. It comprises 19 items yielding seven component scores (subjective sleep quality, latency, duration, efficiency, disturbances, use of sleep medication, and daytime dysfunction). Higher total scores indicate poorer sleep quality.
Generalized Anxiety Disorder Scale (GAD-2) | Baseline, Day 14, and Day 30
  The GAD-2 will assess anxiety symptoms over the past two weeks. Each of the two items is rated from 0 ("not at all") to 3 ("nearly every day"). The total score ranges from 0 to 6, with higher scores indicating greater anxiety. A score ≥3 suggests clinically significant anxiety.
Patient Health Questionnaire-2 (PHQ-2) | Baseline, Day 14, and Day 30
  The PHQ-2 will measure depressive symptoms over the past two weeks. Each of the two items is rated from 0 ("not at all") to 3 ("nearly every day"). The total score ranges from 0 to 6, with higher scores indicating greater depressive symptoms. A score ≥3 suggests clinically significant depression.
Patient Global Impression of Change (PGIC) | Day 14, and Day 30
  The PGIC will assess the participant's overall perception of improvement since starting the intervention. It is rated on a 7-point Likert scale from 1 ("very much improved") to 7 ("very much worse"), with lower scores representing greater perceived improvement.

OTHER OUTCOMES:
System Usability Scale (SUS) | Day 30
  The System Usability Scale (SUS) will be used to evaluate participants' perceived usability and satisfaction with the Fudan Tinnitus Doctor (FTD) conversational AI system at Day 30. The SUS is a 10-item questionnaire rated on a 5-point scale. The total score will be calculated as (sum of adjusted item scores × 2.5), ranging from 0 to 100, with higher scores indicating greater usability.
Net Promoter Score (NPS) | Day 30
  The Net Promoter Score (NPS) will be used to assess participants' likelihood of recommending the Fudan Tinnitus Doctor system to others at Day 30. Participants will rate their likelihood on a scale from 0 (not at all likely) to 10 (extremely likely).
User Engagement Metrics | Continuous during 30-day intervention period
  System usage data will be automatically recorded to assess user adherence and engagement with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Shan Sun, Ph.D, Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Fudan University Eye Ear Nose and Throat Hospital, Otorhinolaryngology Department, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Deidentified individual participant data (IPD) collected for this trial, including outcome measures and baseline characteristics, will be made available upon reasonable request to qualified researchers. Data sharing will require prior approval from the Institutional Review Board of the Eye & ENT Hospital of Fudan University. The DeepSeek-R1 671B model used to support the intervention is open-source and publicly accessible at https://github.com/deepseek-ai/DeepSeek-R1.